CLINICAL TRIAL: NCT05285423
Title: To Evaluate a New Approach of Vocal Cord Lateralization Using Prolene Suture With Prolene Mesh Stabilization
Brief Title: A Novel Approach for VC Lateralization, With Prolene Suture Stabilized Over Prolene Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Muhammad Rashid, Muhammad Rashid, Head of The Department Otolaryngology, Kharian, The Principal Investigator., Pak Emirates Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prolene VC Lateralization
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Paralysis of Vocal Cords or Larynx; Bilateral Vocal Cord Paralysis
Keywords: Voice Rehabilitation; Vocal cord lateralisation; Prolene mesh implant; Bil abductor Vocal Cord Paralysis
MeSH Terms: conditions — Vocal Cord Paralysis; Laryngeal Diseases

STUDY DESIGN:
Intervention Model Description: The single group will be offered vocal cord lateralization with prolene suture and mesh implant technique.
Masking Description: Patients in othe only arm are provided with vocal cord lateralization with prolene suture technique, and this is known by the patient, health care provider and the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolene suture technique. (Experimental): The Group of Patients who were offered Vocal Cord Lateralization with prolene suture technique.
  Interventions: Procedure: Novel technique of Vocal cord Laterlization with Prolene suture.

INTERVENTIONS:
Procedure: Novel technique of Vocal cord Laterlization with Prolene suture. — The procedure will be performed under General anesthesia, preferably with a tracheostomy so that the extent of vocal cord lateralization could be ascertained intraoperatively.

SUMMARY:
The larynx performs important functions of the aero-digestive tract, it has a vital role in the control of breathing, phonation, deglutition, and protection of the lower respiratory tract from aspiration. Bilateral Vocal cord paralysis is a challenging and at times debilitating laryngeal dysfunction that has a great social and economic impact on a patient's life. VC Lateralization, if done accurately and up to the expectations of the patient is very rewarding. However different surgical procedures which include cordectomy, arytenoidectomy with or without laser, open surgical methods, and Isshiki type 2 thyroplasty are in practice. Each has its own profile of benefits and disadvantages. Most of them are technically difficult and complex, need specialized equipment, and are out of reach of the general ENT surgeons. The investigator suggests using the Prolene suture stabilized over Prolene mesh for Vocal Cord Lateralization.

DETAILED DESCRIPTION:
Introduction: The larynx performs important functions of the aero-digestive tract, it has vital role in the control of breathing, phonation, deglutition, and protection of the lower respiratory tract from aspiration. The function of the vocal cord is central to all the Laryngeal functions, even unilateral paralysis can have a profound effect on overall laryngeal functionality especially in sound production. Around 80% of all the jobs in the world are somehow dependent upon social communication. bilateral vocal cord paralysis is a debilitating laryngeal dysfunction that has a great social and economic impact on a patient's life. Lateralization thyroplasty (LT), if done accurately and up to the expectations of the patient is very rewarding. However different surgical procedures which include both endoscopic cordectomy, arytenoidectomy with or without laser, and open surgical methods including Isshiki type 2 thyroplasty are in practice. Each method has its own profile of benefits and disadvantages. Most of them are technically difficult and complex, need specialized equipment, and are out of reach of the general ENT surgeons and population. In this regard, the intended aim is to test a prolene suture stabilized over prolene mesh to lateralize the vocal cord. The Investigator recommends some modifications in the original technique, which would not require complex measurements and costly equipment. Prolene is already in use in a wide range of procedures worldwide, approved by the Federal drug administration in 1997 but it has never been used in the larynx. The objective of this study is to to explore the efficacy of the prolene suture technique with prolene mesh stabilization for vocal cord Lateralization in terms of patient satisfaction and voice outcome.

Objective: To evaluate a new approach of vocal cord Lateralization using prolene suture and mesh.

Study Design: Interventional, prospective study. Place and Duration of study: Ent departments of multiple tertiary care hospitals of Pakistan from Jan 2022 to May 2022.

Materials and Methods: Hospital ethical committee's approval will be obtained. Patients of age 15 years onwards, with bilateral vocal cord paralysis/ paresis due to trauma and idiopathic causes will be included. Patients with neoplasm and underlying muscular dystrophy are to be excluded from the study. All patients will be counseled properly and given the choice of intervention by prolene Suture technique. Consenting patients will be subjected to routine blood investigations, fiber optic laryngoscopy, and imaging with a Computerized Tomography scan (where applicable). The surgery will be performed under General anesthesia. Tracheostomy is preferred to get an adequate view of the glottis and to ascertain the extent of lateralization intraoperatively. The incision will be made at the lower border of thyroid cartilage under aseptic measures. Skin flaps will be raised in the sub-platysmal plane, strap muscles will be separated in the midline to expose the laryngeal cartilaginous framework. Two wide bore Canula (16G) are passed at the levels just above and below the true Vocal cord under laryngoscopic guidance. Prolene 1-0 suture (thickness 0.3-0.4mm) thread is passed through the lower cannula and the thread end is brought out through the upper cannula bore under microscopic forceps guidance. Both the ends are now tied over the thyroid lamina with a prolene mesh between the knot and the cartilage. the tension of the knot determines the extent of lateralization needed. Wound will be closed in layers. The patient will be kept in hospital for a day or more for observation. The success of the surgical procedure will be measured in terms of post-operative decannulation of tracheostomy and preservation of reasonable postop voice with comfortable breathing altogether. Tracheostomy decannulation will be done between 24 to 48 hours post operatively. Preoperatively Voice and breathing parameters will be noted and Post operatively evaluated at day 14. For subjective evaluation of ease of breathing, pre and postoperative Visual Analog score (VASb) will be recorded at Rest and light exercise, graded from 1-10 (1 being the comfortable easy breathing and 10 being the most difficult). Peak expiratory flow (PEF) will be measured for an objective assessment of ease in breathing both pre and post operatively. For subjective assessment of voice quality, Visual analog score (VASV) (1-10) will be used both pre and postoperatively. It will be graded as 1 being the best voice and 10 the worse. For an objective assessment of the patient's voice, a customized Voice Handicap Index (VHI-10) will be used.

Modified VHI-10 Questionnaire:

My voice makes it difficult for people to hear me. 0 1 2 3 4 5

I run out of air when I talk. 0 1 2 3 4 5

People have difficulty understanding me in a noisy room. 0 1 2 3 4 5

I use a great deal of effort to speak. 0 1 2 3 4 5

My family has difficulty hearing me when I call them throughout the house. 0 1 2 3 4 5

I use my phone less often than I would like to. 0 1 2 3 4 5

I am tense when I am talking to others because of my voice. 0 1 2 3 4 5

I tend to avoid groups of people because of my voice. 0 1 2 3 4 5

People seem irritated with my voice. 0 1 2 3 4 5

People ask what's wrong with my voice. 0 1 2 3 4 5

VHI : Voice Handicap Index 0 = never, 1 = almost never (occasionally), 2 = sometimes, 3 = almost always, 4 = always

Modified Voice Handicap Index (VHI-10)

Routine monthly follow-up for 3 months will be advised after that.

The results will be analyzed using International IBM SPSS Statistics version 20. Variables defined would be compared between the preoperative and postoperative groups. For normal data paired sample t-test would be used and for abnormally distributed data nonparametric t-test would be used. A P-value of less than 0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

15 years and above. Vocal cord paralysis

Exclusion Criteria:

Neoplasia Muscular dystrophy trauma Cardiac decompensation Dysfunctional pulmonary variables-

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Decannulation with comfortable breathing and reasonable voice | 14th Postoperative day
  Successful decannulation of the tracheostomy tube and normal breathing pattern without tracheostomy. (Yes/No)
Change in Voice Quality on Visual Analogue Score | Preoperative and 14th Postoperative day
  For subjective assessment of voice quality Visual (1-10) analogue score (VASV) will be used both pre and postoperatively. Score 1 being the best voice and 10 the worse.
Modified VHI-10 Questionnaire | Preoperative and 14th Postoperative day
  My voice makes it difficult for people to hear me. 0 1 2 3 4 5 I run out of air when I talk. 0 1 2 3 4 5 People have difficulty understanding me in noisy room. 0 1 2 3 4 5 I use a great deal of effort to speak. 0 1 2 3 4 5 My family has difficulty hearing me when I call them throughout the house. 0 1 2 3 4 5 I use phone less often than I would like to. 0 1 2 3 4 5 I am tense when I am talking to others because of my voice. 0 1 2 3 4 5 I tend to avoid groups of people because of my voice. 0 1 2 3 4 5 People seem irritated with my voice. 0 1 2 3 4 5 People ask what's wrong with my voice. 0 1 2 3 4 5 VHI : Voice Handicap Index 0 = never, 1 = almost never (occasionally), 2 = sometimes, 3 = almost always, 4 = always Fig 1.1 Modified Voice Handicap Index (VHI-10)
Change in breathing effort on Visual Analogue Score | Preoperative and 14th Postoperative day
  For subjective assessment of voice quality Visual analogue score (VASb) will be used both pre and postoperatively. Score 1 being the comfortable easy breathing and 10 being the most difficult.
Peak Expiratory flow during Rest and Light Exercise, | Preoperative and 14th Postoperative day
  Objective assessment of Ease of breathing during rest and Light exercise. (Ltrs/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad N Karim, FCPS, Principal Investigator — CMH Sialkot
Locations (1):
- ENT Departments, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No